CLINICAL TRIAL: NCT00234624
Title: Hepatic Hemodynamic Changes and Simulation Before /After Living-Related Liver Transplantation in Donors/Recipients
Brief Title: Hepatic Hemodynamic Changes and Simulation in Living-Related Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700821
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2005-10-07 (Estimated); Status verified 2005-09

CONDITIONS: Right Hepatectomy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This 1-year project is intended to study the hemodynamic changes of poratal and hepatic artery during living related liver transplantation. We hypothesize that after right hepatectomy for living related liver transplatation, portal vein overflow will change the remnant liver contour and result in liver hyperplasia.

DETAILED DESCRIPTION:
We use CT as tools to reconstruct 3D images of portal vein and hepatic artery before and one month after operation. The images are transferred to CAD and computer simulation is performed.

ELIGIBILITY:
Inclusion Criteria: - Informed adult-to adult living donor underwent right lobectomy

Exclusion Criteria:

* no written informed contents

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Po-Huang Lee, PhD, Principal Investigator — NTUH
Locations (1):
- NTUH, Taipei, Taiwan